CLINICAL TRIAL: NCT00133653
Title: The Impact of Job Strain and Marital Cohesion on Ambulatory Blood Pressure Over One Year: The Double Exposure Study
Brief Title: The Double Exposure Study: The Impact of Job Strain and Marital Cohesion on Blood Pressure
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: DE-2001
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2005-10-31 (Estimated); Status verified 2004-08

CONDITIONS: Hypertension
Keywords: Hypertension; Job Strain; Marital Strain; Blood Pressure
MeSH Terms: conditions — Hypertension; Occupational Stress | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Observational

SUMMARY:
Psychosocial and lifestyle stressors, such as job strain (JS) and marital factors have previously been associated with a sustained increase in blood pressure (BP).

In a one-year longitudinal follow-up to the Baseline Double Exposure cohort study, we, the researchers at Sunnybrook and Women's College Health Sciences Centre, evaluated whether JS and marital cohesion continued to be associated with ambulatory blood pressure (ABP) in subjects enrolled with normal or untreated high BP.

DETAILED DESCRIPTION:
Psychosocial and lifestyle stressors, such as job strain (JS) and marital factors have previously been associated with a sustained increase in blood pressure (BP).

In a one-year longitudinal follow-up to the Baseline Double Exposure cohort study, we evaluated whether JS and marital cohesion continued to be associated with ambulatory blood pressure (ABP) in subjects enrolled with normal or untreated high BP.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65
* Unmedicated for at least 6 months
* Living with spouse for at least 6 months
* Working for at least 6 months

Exclusion Criteria:

* Working rotating or evening shifts

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2001-08; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon W Tobe, MD, Principal Investigator — Sunnybrook & Women's College Health Sciences Centre
Locations (1):
- Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Baker B, Paquette M, Szalai JP, Driver H, Perger T, Helmers K, O'Kelly B, Tobe S. The influence of marital adjustment on 3-year left ventricular mass and ambulatory blood pressure in mild hypertension. Arch Intern Med. 2000 Dec 11-25;160(22):3453-8. doi: 10.1001/archinte.160.22.3453. PMID 11112239